CLINICAL TRIAL: NCT05002582
Title: Carbapenem-resistant Organisms (CRO) Screening From Rectal Swabs and the Relationship Between Colonization and Infection in Patients With Hematological Diseases in China
Brief Title: Carbapenem-resistant Organisms (CRO) Screening From Rectal Swabs in Patients With Hematological Diseases in China
Acronym: CROSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Jian-cang Zhou M.D., Professor, Sir Run Run Shaw Hospital
Other Study IDs: SRRSH-CROSS
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Hematological Diseases; Carbapenem-resistant Enterobacteriaceae; Carbapenem-resistant Pseudomonas Aeruginosa; Carbapenem-resistant Acinetobacter Baumannii
Keywords: Carbapenem-resistant Organisms; colonization; hematological diseases; rectal swabs
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with hematological diseases: to clarify the intestinal carriage rate of carbapenem-resistant Organisms (CRO) in patients with hematological diseases

SUMMARY:
Carbapenem-resistant Organisms (CRO) include Carbapenem-resistant Enterobacteriaceae (CRE), Carbapenem-resistant Pseudomonas aeruginosa (CRPA) and Carbapenem-resistant Acinetobacter baumannii (CRAB). Due to the high fatality rate of CRO infection, and its potential for wide spread, it is currently one of the issues that seriously affect the global public health safety. In 2019, CDC of the United States listed CRE and CRAB as the highest level of "antibiotic-resistant bacteria with urgent threat", while CRPA was listed as "antibiotic-resistant bacteria with serious threat".

Previous studies show that in China, patients with hematological disease are at high-risk of CRE colonization and infection, but there still lack the data of colonization rate of CRPA and CRAB in patients with hematological disease. Intestinal flora is not only an important micro-ecological environment for the human body, but also an important place for the habitation of multidrug-resistant bacteria. The colonization of these bacteria can not only lead to the spread of bacteria in hospital, but also may lead to the translocation infection of carriers. Patients with hematological diseases are often in a state of neutropenia after chemotherapy. At the same time, chemotherapy drugs and various factors can cause intestinal mucosa damage, which is prone to induce intestinal microflora translocation, causing serious infections such as sepsis, and posing a serious threat to the prognosis of patients. Early detection of CRO carriers is not only beneficial to the control of nosocomial infection, but also beneficial to early precise anti-infection treatments, reducing the probability of infection and improving the prognosis of infected patients.

Our study is designed to clarify the intestinal carriage rate of carbapenem-resistant Organisms (CRO) in patients with hematological diseases, and the risk factors of intestinal CRO colonization in patients with hematological diseases and its correlation with subsequent infections. 5000 patients diagnosed with hematological diseases will be enrolled, and rectal swabs or feces will be collected to detect the CRE intestinal colonization. Subsequently, the last 6 months clinical data of CRO-colonized patients and matched non CRO-colonized patients (1:1) will be collected. Then, the randomly selected 200 CRO-colonized patients and matched 200 non CRO-colonized patients (1:1) are followed up for 12 months, a total of 400 patients will be enrolled. Every month, rectal swabs and relevant clinical data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* On a certain day in each chosed hospital, all the inpatients diagnosed with hematological malignancies diseases will be enrolled

Exclusion Criteria:

* Patients or their legal representatives refused to enter the study
* Patients died because of hematological malignancies diseases.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study focused on the colonization rate of Carbapenem-resistant Organisms (CRO) in the intestine of Chinese patients with hematological malignancies diseases, who are at high-risk of CRE colonization and infection, but there still lack the data of colonization rate of CRPA and CRAB in patients with hematological disease.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
CRO intestinal colonization incidence | 1 year since enrollment
  Positive culture any of these three organsisms: Carbapenem-resistant Enterobacteriaceae (CRE), Carbapenem-resistant Pseudomonas aeruginosa (CRPA) and Carbapenem-resistant Acinetobacter baumannii (CRAB)

SECONDARY OUTCOMES:
Bloodstream infection incidence | 1 year after enrollment
  Blood postive culture of the same organisms found in the rectal swabs

CONTACTS AND LOCATIONS:
Overall Officials: Yunsong YU, MD, Principal Investigator — Zhejiang University school of medicine
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu H, Huang W, Ruan S, Zhou J, Wang Y, Weng R, Shi Q, Jiang Y, Jin X, Yu Y. Intestinal colonization of carbapenem-resistant gram-negative bacteria in pediatric hematology patients: risk factors and molecular characteristics, a multicenter case-control study. BMC Microbiol. 2025 Dec 17;25(1):794. doi: 10.1186/s12866-025-04533-z. PMID 41408155
- [Derived] Hu H, Wang Y, Sun J, Wang Y, Zhou J, Shi Q, Han X, Jiang Y, Wu D, Huang X, Yu Y. Risk factors and molecular epidemiology of intestinal colonization by carbapenem-resistant Gram-negative bacteria in patients with hematological diseases: a multicenter case-control study. Microbiol Spectr. 2024 Jul 2;12(7):e0429923. doi: 10.1128/spectrum.04299-23. Epub 2024 Jun 7. PMID 38847538